CLINICAL TRIAL: NCT05544136
Title: A Pilot Study of Radiation De-Escalation for p16 Negative Oropharyngeal Cancer and p16-Negative or Positive Laryngeal and Hypopharyngeal Cancers
Brief Title: A Study of Decreasing Radiation Therapy and Chemotherapy in People With Head and Neck Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-227
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Cancer; Head and Neck Carcinoma; Head and Neck Neoplasms; Head and Neck Squamous Cell Carcinoma
Keywords: Unknown Primary Squamous Cell Carcinoma; Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; fluoromisonidazole; 18F-FMISO; Memorial Sloan Kettering Cancer Center; 22-227
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Neoadjuvant Therapy; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Participants with Squamous Cell Carcinoma Head and Neck Cancer (Experimental): Participants will be hypoxia-negative T0-3N1-2B small cell carcinoma head and neck cancer/SCC HNC patients (HPV-OPC, HPV- UPC with nodal metastasis(es), HPC, or LXC) who are eligible for definitive CRT with de-escalated radiation concurrent with 2 cycles of SOC chemotherapy. Hypoxia status will be determined by the absence of hypoxia radiotracer uptake on 18F-FMISO PET/CT imaging
  Interventions: Diagnostic Test: 18F-FMISO PET/CT scan; Radiation: Chemoradiation therapy; Drug: Carboplatin

INTERVENTIONS:
Diagnostic Test: 18F-FMISO PET/CT scan — 18F-FMISO PET/CT scan (only 1 injection) that occurs 5-10 treatment days after RT start
Radiation: Chemoradiation therapy — * 18F-FMISO hypoxia negative patients complete CRT with 70Gy primary tumor and 50Gy de-escalated RT dose to gross nodes (if 50Gy is has pilot efficacy, then 44Gy to gross nodes; if 44Gy has pilot efficacy, then 40Gy to gross nodes).
  * 18F-FMISO hypoxia positive patients are taken off study and complete SOC 70Gy CRT to primary tumor and gross nodes.
  Other Names: CRT
Drug: Carboplatin — The chemotherapy used in this protocol is the standard of care for head and neck cancer, cisplatin or carboplatin/5-Fluorouracil

SUMMARY:
The purpose of this study is to test the treatment approach of de-escalated radiation and chemotherapy followed by a planned neck dissection surgery in people with head and neck cancer. The study will look at how effective the treatment approach is against participants' cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of SCC of the head and neck (excluding nasopharynx, nasal cavity/paranasal sinus, oral cavity, salivary, thyroid, and cutaneous primary malignancies).

  * Any unknown primary SCC of the head and neck with radiographically detectable gross nodes is allowed (core or excisional biopsy acceptable; if excisional biopsy is performed, there must be residual radiographically detectable nodal disease; FNA may be acceptable only with PI and/or co-PI approval)
  * If the primary site is oropharynx or unknown primary, P16 IHC must be negative.
  * If the primary site is hypopharynx or larynx, any P16 status is acceptable (positive, negative, or unknown). P16 IHC is strongly encouraged when possible.
* Clinical stage T0-3 N1-2C M0 (AJCC 7th edition) without evidence of distant metastasis based on staging FDG PET/CT.
* 18 years of age or older.
* Must not have received prior radiation therapy or chemotherapy for HNC.
* Patients who have had their primary site tumor removed by surgery but still have residual grossly enlarged, radiographically detectable lymph nodes are eligible for this study.
* Karnofsky Performance Status (KPS) ≥ 70.
* CT or MRI of the Neck with and without contrast

  o Note: A CT scan of the Neck and/or a PET/CT performed for the purposes of radiation planning may serve as planning tools.
* Adequate hematologic function within 30 days prior to registration, defined as follows:

  * White Blood Count (WBC) ≥ 2,000 cells/µL
  * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3
  * Platelets ≥ 100,000 cells/mm3
  * Hemoglobin ≥ 8.0 g/dL; Note: The use of transfusion or other interventions to achieve Hgb ≥ 8.0 g/dL is acceptable
* Adequate renal function within 30 days prior to registration, defined as follows:

  * Serum creatinine < 1.5 mg/dL or creatinine clearance (CrCl) ≥ 50 mL/min determined by 24-hour collection or estimated by Cockcroft-Gault formula: CrCl male = [(140 - age) x (weight in kg)] / [(Serum Cr mg/dL) x (72)] CrCl female = 0.85 x (CrCl male)
  * Patients with serum creatinine > 1.5 mg/dL can be eligible for carboplatin-based chemotherapy with approval of co-PI (Dr. Eric Sherman
* Adequate hepatic function within 30 days prior to registration, defined as follows:

  * Bilirubin < 2 mg/dL
  * AST or ALT < 3 x the upper limit of normal
* Negative serum pregnancy test within 14 days prior to registration for women of childbearing potential.
* The subject/legally authorized representative (LAR) must provide study-specific informed consent prior to study entry.

Exclusion Criteria:

* All nasopharyngeal, nasal cavity/paranasal sinus, oral cavity, salivary gland, thyroid, and cutaneous primary malignancies.
* Any T4 or N3 patients
* Any prior radiotherapy to the head and neck region.
* Any prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different non-H&N cancer is permissible.
* Prior chemotherapy or radiotherapy within the last three years.
* Patients who underwent previous surgical resection for the same disease (except for biopsy or surgery removing primary site tumor but still present with grossly enlarged, radiographically detectable lymph nodes).
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for 3 years or if cure rate from treatment at 5 years estimated to be ≥ 90%.
* Subjects with simultaneous primary cancers outside of the oropharynx

  o Note: Exceptions can be made for patients with simultaneous primaries outside the H&N if determined by the PI/Co-PI that the patient can proceed with protocol activities.
* Pregnant (confirmed by serum b-HCG in women of reproductive age) or breastfeeding.
* Severe, active co-morbidities defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months.
  * Transmural myocardial infarction within the last 6 months.
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration.
  * Hepatic Insufficiency resulting in clinical jaundice and/or coagulation defects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2027-03-12 (Estimated); Study Completion 2027-03-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants alive post-Chemo Radiation Therapy | 2.5 years
  The primary objective is to assess the pilot efficacy of RT dose de-escalation to grossly involved lymph nodes for hypoxia negative T0-T3N1-2B HPV- OPC/UPC and HPC/LXC patients. For evaluation on the efficacy of the regimen in this cohort, a simple decision rule will be implemented as follows: If, among the first 10 evaluable patients, we have at least 8 patients who are alive, followed, and have major pathological response on planned neck dissection at 4 months ± 1 month post-CRT, then we will declare the treatment modality using that RT dose has pilot efficacy and will then proceed with treatment at the next de-escalated dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab Abou Yehia, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org